CLINICAL TRIAL: NCT05839652
Title: Treatment of Orthostatic Hypotension in Individuals With Spinal Cord Injury
Brief Title: Treatment of Orthostatic Hypotension in SCI
Acronym: SCI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Scientist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1747301-1
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Midodrine; Droxidopa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study 1 (Experimental): Twenty-five participants will be asked to visit the laboratory on 6 occasions, for an open-label, dose escalation trial to determine the effect of midodrine and droxidopa on supine and seated blood pressure and on symptoms of autonomic dysreflexia and orthostatic hypotension.
  Interventions: Drug: Midodrine Hydrochloride
- Study 2 (Experimental): Determine the effects of compression garments, midodrine, and droxidopa, compared to placebo, on orthostatic hemodynamics, symptoms of AD and OH and reporting of fatigue and thermal comfort.
  Interventions: Drug: Midodrine Hydrochloride

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Determine best drug and dose to increase and stabilize SBP during orthostatic tilt
  Other Names: Droxidopa

SUMMARY:
The purpose of this study is to identify the effects of non-pharmacological and pharmacological anti-hypotensive treatment interventions on orthostatic hemodynamic responses, symptoms of autonomic dysreflexia and orthostatic hypotension, and levels of fatigue and comfort in hypotensive individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord injury
* at least 12 months post injury
* injury level of C1-T6
* AIS A, B or C
* non-ambulatory
* non-ventilator

Exclusion Criteria:

* Active psychiatric disorder
* Stroke or cerebrovascular disease
* Alzheimer's Disease or dementia
* Unmanaged cardiac arrhythmias
* Concurrent systemic, hepatic, or renal disease
* Suspected or diagnosed malignancy
* Neurological disease other than SCI
* Self-reported history of three or more symptomatic episodes of AD per day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 years
  determine differences in systolic blood pressure after midodrine, droxidopa, compression stockings and placebo

SECONDARY OUTCOMES:
Cerebral blood flow velocity | 3 years
  determine differences in cerebral blood flow velocity after midodrine, droxidopa, compression stockings and placebo
Symptoms of autonomic dysreflexia and orthostatic hypotension | 3 years
  determine differences in symptoms after midodrine, droxidopa, compression stockings and placebo

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kessler Foundation, West Orange, New Jersey
  - James J Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No